CLINICAL TRIAL: NCT00204919
Title: Intermittent Vitamin D Administration in the Nursing Home: Impact on Vitamin D Status, Falls, Bone Turnover and Bone Density
Brief Title: Vitamin D Administration in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001-099
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2015-09

CONDITIONS: Vitamin D Deficiency; Osteoporosis
Keywords: osteoporosis; vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis | interventions — Vitamin D; Ergocalciferols; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Active Comparator)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — once-monthly vitamin D oral capsules (50,000 units)
  Other Names: ergocalciferol
  Arms: 2
Drug: placebo — once-monthly placebo capsules
  Other Names: lactose
  Arms: 1

SUMMARY:
Administration of vitamin D 50,000 units once monthly will:

* Maintain serum 25-OH vitamin D above 20 ng/ml
* Reduce falls
* Increase calcaneal BMD
* Reduce bone turnover
* Be well tolerated: volunteers will not develop hypercalcemia
* Improve performance on a swallowing quality of life questionnaire

DETAILED DESCRIPTION:
1. Research questions: We propose a prospective double-blind, randomized, placebo-controlled trial of once-monthly vitamin D oral capsules (50,000 units) in nursing-home residents.

Subjects from several Wisconsin nursing homes were randomized to receive once-monthly vitamin D oral capsules (50,000 units) or placebo. Blood levels of 25-OH D, parathyroid hormone, serum calcium, and a marker of bone turnover will be measured periodically by standard lab assays. Swallowing quality of life was measured by questionnaire. Appropriate statistical tests (paired T tests, 95% confidence intervals will be calculated with the large sample approximation for binomial variables, other).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Nursing Home Resident in Wisconsin

Exclusion Criteria:

* Renal Failure
* Hypercalcemia
* Metastatic Cancer

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2001-06; Primary Completion 2004-05 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Plasma 25-hydroxyvitamin D levels | 1 year

SECONDARY OUTCOMES:
Plasma calcium | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elliott, PharmD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States